CLINICAL TRIAL: NCT06938906
Title: Survival Outcome Analysis on the Strategy Shift Integrating a Multimodal Therapy of Neoadjuvant Chemotherapy and Extended Pancreatectomy in Pancreatic Cancer: A Clinical Study From a Retrospective Cohort in a Single Institute
Brief Title: Multimodal Therapy Impact on Pancreatic Cancer Survival
Acronym: MMTIPS
Status: Active, not recruiting | Type: Observational
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Ting-Kai Liao, Principal Investigator, Director of Specialized Ward for Division of General Surgery, Department of Surgery, National Cheng Kung University
Other Study IDs: NCKUH-11405009
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer; Neoadjuvant Chemotherapy; Pancreatectomy
Keywords: pancreatic cancer; neoadjuvant chemotherapy; extended pancreatectomy; multimodal therapy; paradigm shift; survival outcomes
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: The patient of pancreatic cancer, who began to have treatment in the period between 2011 to 2017.
- Group B: The patient of pancreatic cancer, who began to have treatment in the period between 2018 to 2022.

SUMMARY:
The goal of this retrospective cohort study is to analyze change of treatment strategies affect the survival outcomes in patients of pancreatic cancer who received curative-intent treatment. The main question it aims to answer is:

Hypothesis: Change of treatment strategies involving increased utility of neoadjuvant chemotherapy and aggressive surgical approaches of extended pancreatectomy improved the overall and progression free survival in the patients with pancreatic cancer.

Participants received curative treatment for pancreatic cancer.

DETAILED DESCRIPTION:
This study is to analyze the change of treatment strategies and shift of the paradigm over time in a single center. Researchers plan to see the impact of the evolvement to the survival outcomes in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic adenocarcinoma
* Received curative surgery

Exclusion Criteria:

* Other subtypes of pancreatic cancer including acinar cell carcinoma, mucinous carcinoma, undifferentiated carcinoma and intraductal papillary mucinous neoplasm with associated adenocarcinoma
* Cases with palliative or R2 resection were also excluded from the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic cancer who lived in southern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2011-01-03 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival and Progression-free survival | From enrollment to two years after the end of treatment
  Overall survival was calculated from the first treatment day of the disease to the day of mortality. Progression-free survival was calculated from the first treatment day of the disease to the day of proression or recurrece of pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Shen Shan, MD., PhD., Study Chair — Department of Surgery, National Cheng Kung University Hospital; Ting-Kai Liao, MD., Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided